CLINICAL TRIAL: NCT01788800
Title: The Influence of Physical Activity on the Effect of Cognitive Behavioural Therapy, Neurobiological Parameters and Information Processing in Patients With Panic Disorder With/Without Agoraphobia
Brief Title: Physical Activity and Cognitive Behavioural Therapy in Panic Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Principal Investigator, Prof. Dr. Andreas Ströhle, Prof. Dr., Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 221012
Record Dates: First submitted 2013-02-04; First posted 2013-02-11 (Estimated); Last update posted 2013-05-16 (Estimated); Status verified 2013-05

CONDITIONS: Panic Disorder
Keywords: Panic disorder; Physical activity
MeSH Terms: conditions — Panic Disorder; Motor Activity | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise training (Experimental): Cognitive Behavioural Therapy (CBT)
  + Exercise training 3 times/week, 30 minutes on a treadmill, 70% maximal oxygen uptake (VO2max), 8 weeks
  Interventions: Behavioral: Cognitive Behavioural Therapy (CBT)
- Movements (Active Comparator): Cognitive Behavioural Therapy (CBT)
  + Low intensity physical activity without cardiovascular activation, 3 times/week, 30 minutes, 8 weeks
  Interventions: Behavioral: Cognitive Behavioural Therapy (CBT)

INTERVENTIONS:
Behavioral: Cognitive Behavioural Therapy (CBT) — 9 sessions of CBT including psychoeducation and interoceptive exposure

SUMMARY:
Physical activity (treadmill) supports the effect of cognitive behavioural therapy in patients with panic disorder with/without agoraphobia

DETAILED DESCRIPTION:
Patients undergo cognitive behavioural therapy consisting of 8 group sessions within 1 month. All patients additionally complete a training of physical activity, which starts simultaneously to therapy and runs for 8 weeks (3 times/week, 30 minutes each). Half of the patients complete training on a treadmill while the other half completes a training programme of low intensity physical activity without cardiovascular activation.

Flanking EEG (electroencephalogram) recordings shall help clarify biological processes underlying the therapeutical process.

ELIGIBILITY:
Inclusion Criteria:

1. Subject familiarized with experimental procedure and had given written informed consent
2. Diagnosis of panic disorder with or without agoraphobia according to Diagnostic and Statistical Manual of Mental Disorders (DSM-IV)
3. Sufficiently able to communicate with investigator, answer questions and fill in questionnaires
4. Reachability of patient for treatment and follow-up

Exclusion Criteria:

1. Other psychiatric illnesses like schizophrenia, substance abuse or severe depressive episode
2. Acute suicidal tendency
3. Epilepsy or other illness of the central nervous system (e.g. brain tumor, encephalitis)
4. Existence of contraindication against physical exercise
5. Pregnancy or breastfeeding
6. Changes of psychopharmacological treatment within the last 4 weeks

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2009-01; Primary Completion 2013-01 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Hamilton Rating Scale for Anxiety (CIPS 1995) | up to 28 weeks (follow up)
  Global interviewer rated measure for anxiety and severity indicator of an anxiety disorder

SECONDARY OUTCOMES:
Panic and Agoraphobia Scale (Bandelow et al. 1995) | Baseline, 4 weeks, 8 weeks and 28 weeks (follow up)
Beck Anxiety Inventory (CIPS 1995) | Baseline, 4 weeks, 8 weeks and 28 weeks (follow up)
Clinical Global Index (CIPS 1995) | Baseline, 4 weeks, 8 weeks and 28 weeks (follow up)
Beck Depression Inventory (CIPS 1995) | Baseline, 4 weeks, 8 weeks and 28 weeks (follow up)

OTHER OUTCOMES:
EEG and endocrinology | Baseline, 4 weeks, 8 weeks and 28 weeks (follow up)
  EEG (Mismatch Negativity, Loudness dependency, P50/P300) and diurnal profile of Cortisol and alpha-Amylase

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Ströhle, Prof. Dr., Principal Investigator — Department of Psychiatry and Psychotherapy, CCM, Charité - Universitätsmedizin Berlin

REFERENCES:
- See also: Related Info — http://www.angstambulanz-charite.de